CLINICAL TRIAL: NCT06766747
Title: Efficacy of Intermittent Fasting Versus Continuous Caloric Restriction in the Treatment of Significant Weight Regain After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-CIE-0622-23
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Obesity Prevention; Bariatric Surgery Complications; Intermittent Fasting
Keywords: Gain Weight Following Bariatric Surgery; Intermittent Fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Masking Description: person in charge of statistical analysis and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Participants in the alternate-day fasting group will receive biweekly telecounseling to ensure adherence to the prescribed dietary plan and to monitor for potential adverse events. During the 12-week weight loss phase, patients are instructed to restrict calories to 75% of usual intake 2 days per week. A daily intake of at least 2 liters of low-energy beverages (water, caffeine- and sugar-free beverages) is generally recommended on fasting days. Usual physical activity is encouraged to continue except on fasting days.
  Interventions: Other: Intermittent Fasting
- Control group (Placebo Comparator): Participants in the continuous calorie restriction group will receive biweekly nutritional counseling via telecoaching to ensure adherence to the prescribed dietary plan. Based on the weekly caloric intake obtained from the 7-day log, a model menu will be prescribed with 25% daily caloric restriction divided into 3 meals per day consisting of macronutrient intake with 20% of energy as fat, 40 to 50% as carbohydrate, and 20 to 30% as protein. They are instructed to continue their usual physical activity.
  Interventions: Other: Continuous calorie restriction

INTERVENTIONS:
Other: Intermittent Fasting — Participants in the alternate-day fasting group will receive biweekly telecounseling to ensure adherence to the prescribed dietary plan and to monitor for potential adverse events. During the 12-week weight loss phase, patients are instructed to restrict calories to 75% of usual intake 2 days per week. A daily intake of at least 2 liters of low-energy beverages (water, caffeine- and sugar-free beverages) is generally recommended on fasting days. Usual physical activity is encourage
  Arms: Intervention group
Other: Continuous calorie restriction — Participants in the continuous calorie restriction group will receive biweekly nutritional counseling via Telecoaching to ensure adherence to the prescribed dietary plan. Based on weekly caloric intake obtained from the 7-day log, a model menu will be prescribed with a 25% daily calorie restriction divided among 3 meals every day consisting of macronutrient intake, with 20% of energy as fat, 40 to 50% as carbohydrate, and 20 to 30% as protein. They will be instructed to continue their usual physical activity.
  Arms: Control group

SUMMARY:
Intermittent fasting has gained relevance in recent years because it allows for significant weight loss with improvement in cardiovascular risk factors similar to calorie-restricted diets without people having to track calories every day, or prohibiting people from eating certain food groups. However, there is no data about its usefulness in patients with weight gain after bariatric surgery, or its long-term effects(9).

Research question: In patients with weight gain, being followed up in the obesity clinic, is intermittent fasting for 12 weeks, compared to calorie restriction, effective in terms of weight reduction?

H0: Change in weight from baseline to 12 weeks less than 5% H1: Change in weight from baseline to 12 weeks greater than or equal to 5%

Patients meeting the inclusion criteria will be identified. Once identified, they will be asked to participate in the study and, if they accept, they will be asked to complete and sign the informed consent form. The study will consist of three phases: a selection phase, an adaptation phase (1 to 2 weeks), a weight loss phase (12 weeks) and a maintenance phase (12 weeks).

At the first visit, patients will be randomized to two types of nutritional interventions: intermittent fasting or caloric restriction. During the weight loss phase, biweekly follow-up will be performed to ensure adherence to the assigned dietary intervention. At the end of the 12 weeks, patients can decide whether to continue the assigned dietary intervention or move to a maintenance plan. Anthropometric measurements and body composition will be measured at baseline, 12 and 24 weeks.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will be identified. Once identified, they will be asked to participate in the study and, if they accept, they will be asked to complete and sign the informed consent form. The study will consist of three phases: a selection phase, an adaptation phase (1 to 2 weeks), a weight loss phase (12 weeks) and a maintenance phase (12 weeks).

Selection Period (Visit 0)

The bariatric surgery, nutrition, and endocrinology consultation of the bariatric clinic will identify possible candidates. In addition, the use of dietary supplements will be reviewed according to the Obesity Clinic's Clinical Practice Guide and the labs necessary to complete the baseline cardiometabolic profile will be obtained. A 7-day food recall and a record of usual physical activity and signing of informed consent will be required. In addition, an application will be downloaded to assess the number of steps per day taken by the individual to control for the physical activity variable.

Adjustment period (visit 1)

A visit with an obesity clinic dietitian will be scheduled 7 to 14 days after selection. During this visit, the 7-day recall will be reviewed to calculate basal weekly caloric intake. Baseline clinical and anthropometric data (weight, height, body mass index, abdominal circumference, and body composition) will be collected. Randomization will then be performed using a simple computer-generated randomization code, which will be managed centrally by a person who is unaware of the clinical characteristics of each patient outside the research group. The allocation made by this mechanism cannot be changed by the treating physicians. Subjects who do not attend the second visit or who do not properly complete the 7-day food and exercise diaries will be excluded. The order for the new metabolic profile will be generated to be performed at the end of the weight loss period.

Weight Loss Period

* Intervention Group (5:2): Participants in the alternate-day fasting group will receive bi-weekly nutritional counseling via telecounseling to ensure adherence to the prescribed dietary plan and to monitor for potential adverse events. During the 12-week weight loss phase, patients will be instructed to restrict their caloric intake to 75% of their usual intake 2 days per week. A daily intake of at least 2 liters of low-energy beverages (water, caffeine- and sugar-free beverages) is generally recommended on fasting days. Usual physical activity is encouraged to continue except on fasting days.
* Control group: Participants in the continuous caloric restriction group will receive biweekly nutritional counseling via telecounseling to ensure adherence to the prescribed dietary plan. Based on the weekly caloric consumption obtained from the 7-day record, a sample menu will be prescribed with a daily caloric restriction of 25%, divided into 3 meals per day, consisting of macronutrient intake with 20% of energy as fat, 40 to 50% as carbohydrate, and 20 to 30% as protein. The patient is instructed to continue normal physical activity.

At the end of the 12-week follow-up, visit 2 (V2) will be scheduled to obtain anthropometric data, body composition, and to review the cardiometabolic profile.

Maintenance period

At visit 2, patients who wish to discontinue intermittent fasting or continuous caloric restriction will be transitioned to a weight maintenance regimen which will be prescribed by a nutritionist from the obesity clinic. In addition, they will be recommended to continue physical activity, verify adherence to dietary supplements, and a follow-up will be scheduled in 12 weeks (visit 3) for anthropometric and cardiovascular profile monitoring.

Alternatively, patients in the intervention group who wish to continue will be prescribed a modified version of fasting. Energy intake on fasting days will be increased from 1000 to 1200 kcal. Similarly, in the continuous caloric restriction group, dietary caloric intake will be increased in a similar proportion. They will be recommended to continue physical activity, verify adherence to dietary supplements, and a follow-up will be scheduled in 12 weeks (visit 3) for anthropometric and cardiovascular profile monitoring.

Final measurements will be taken at week 24, after the two follow-up periods, so that all patients have the measurement at the same intervention time.

ELIGIBILITY:
Patients between 18 and 69 years of age treated with primary and/or secondary bariatric surgery with more than 1 year of postoperative.

2.3.3 INCLUSION CRITERIA

* 10% weight gain with respect to the minimum postoperative weight and/or
* Weight gain rate ≥0.50% with respect to previous weight.
* Supplementation with ferrous sulfate, cyanocobalamin and cholecalciferol, according to clinical criteria.
* Not having modified the therapy in the last 3 months
* Access to mobile phone with data.
* Agree to participate in the study including signing informed consent.

2.3.4 EXCLUSION CRITERIA.

* Patient diagnosed with type 1 diabetes mellitus.
* Patient diagnosed with type 2 diabetes mellitus treated with insulin.
* History of an eating disorder such as anorexia or bulimia. • Untreated vitamin B12, iron, calcium, and/or vitamin D deficiency.
* History of hospitalization for cardiovascular disease (angina, myocardial infarction, or stroke) 3 months prior to the study.
* Use of antidepressant or anti-anxiety medications
* Use of medications that affect the results of the study (weight loss medications)
* Unable to keep a food diary or activity log for 7 consecutive days during screening
* Cognitive impairment that, in the opinion of the principal investigator or study physician, would result in failure to cooperate with study procedures.
* Active neoplastic disease.
* Pregnancy or breast-feeding, or planning to become pregnant during the study period
* Significant psychiatric illness, kidney disease, severe liver disease, or other illness that affects the ability to complete the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Weight loss (Kg) | 12 weeks
  To evaluate the efficacy of intermittent fasting (5:2 diet) for 12 weeks, compared with continuous caloric restriction, in terms of weight reduction in kilograms (Kg), in patients with weight regain.

SECONDARY OUTCOMES:
Percentage of fat mass | 12 weeks
  To describe the change in percentage of fat mass measured at baseline and at 12 weeks of follow-up using the Seca mBCA 554 Medical Body Composition Analyzer.
Visceral fat | 12 weeks
  To describe the change in visceral fat (VAT) measured at baseline and at 12 weeks of follow-up using the Seca mBCA 554 Medical Body Composition Analyzer.
Percentage of lean mass | 12 weeks
  To describe the change in body composition percentage of lean mass measured at baseline and at 12 weeks of follow-up using the Seca mBCA 554 Medical Body Composition Analyzer.
HbA1c | 12 weeks
  Compare changes in HbA1c after 12 weeks of follow-up between the intermittent fasting group and the continuous calorie restriction group.
Weight 24 weeks | 24 weeks
  Compare changes in weight in kilograms after 24 weeks of follow-up.
Percentage of fat mass 24 weeks | 24 weeks
  To describe the change in percentage of fat mass measured at baseline and at 24 weeks of follow-up using the Seca mBCA 554 Medical Body Composition Analyzer.
Visceral fat 24 weeks | 24 weeks
  To describe the change in visceral fat (VAT) measured at baseline and at 24 weeks of follow-up using the Seca mBCA 554 Medical Body Composition Analyzer.
Percentage of lean mass 24 weeks | 24 weeks
  To describe the change in body composition percentage of lean mass measured at baseline and at 24 weeks of follow-up using the Seca mBCA 554 Medical Body Composition Analyzer.
HbA1c 24 weeks | 24 weeks
  Compare changes in HbA1c after 24 weeks of follow-up between the intermittent fasting group and the continuous calorie restriction group.

CONTACTS AND LOCATIONS:
Overall Officials: Diana C Henao, Endocrinologyst, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital Universitario San Ignacio., Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes
The data are available from the authors if requested by the reader for research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code